CLINICAL TRIAL: NCT07100951
Title: Comparing the Efficacy of Brief Psychoanalytic Couple Therapy and Emotionally Focused Therapy in Reducing Relationship Distress and Psychopathological Symptoms: A Randomized Controlled Trial
Brief Title: Comparing Brief Psychoanalytic Couple Therapy and Emotionally Focused Therapy in Reducing Relationship Distress
Acronym: BPCT-EFT-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Istanbul Nisantasi University (Other); Uskudar University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Principal Investigator, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPCT_vs_EFT_RCT_2025
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Depressive Disorder; Anxiety Disorders; Emotion Regulation; Attachment; Relationship Distress
Keywords: Brief Psychoanalytic Couple Therapy; Emotionally Focused Therapy; Couple Therapy; Online Psychotherapy; Relationship Distress; Emotion Regulation; Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Emotional Regulation; Depression | interventions — Emotion-Focused Therapy

STUDY DESIGN:
Intervention Model Description: Participants (60 couples) will be randomly assigned in equal numbers to one of three parallel groups: Brief Psychoanalytic Couple Therapy (BPCT), Emotionally Focused Therapy (EFT), or a Waitlist Control group. Each active therapy group will receive 12 weekly online sessions. Assessments will be conducted at baseline, mid-treatment, post-treatment, and 6-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Psychoanalytic Couple Therapy (BPCT) (Experimental): Couples in this arm will receive 12 weekly online sessions (50 minutes each) of Brief Psychoanalytic Couple Therapy (BPCT). Therapy focuses on unconscious relational dynamics, early attachment schemas, and projective identification. The therapist facilitates insight through interpretation of symbolic meaning in conflict and reenactments of early object relations. The stance is neutral and exploratory.
  Interventions: Behavioral: Brief Psychoanalytic Couple Therapy
- Emotionally Focused Therapy (EFT) (Active Comparator): Couples in this arm will receive 12 weekly online sessions (50 minutes each) of Emotionally Focused Therapy (EFT). EFT targets negative emotional interaction cycles, encourages expression of primary emotions, and fosters attachment security. The therapist plays an active and emotionally attuned role to restructure relational bonds and increase responsiveness between partners.
  Interventions: Behavioral: Emotionally Focused Therapy
- Waitlist Control (No Intervention): Couples in the waitlist control group will not receive active intervention during the 12-week study period but will complete the same assessments at all time points. After the 6-month follow-up assessment, they will be offered a choice of therapy (BPCT or EFT) outside the study protocol.

INTERVENTIONS:
Behavioral: Brief Psychoanalytic Couple Therapy — Brief Psychoanalytic Couple Therapy (BPCT) consists of 12 weekly online sessions (50 minutes each) focused on uncovering unconscious relational dynamics, symbolic conflict meanings, and early attachment schemas. Techniques include relational interpretations, exploration of projective identification and transference, and analysis of emotional defenses. Therapists maintain a neutral, reflective stance to promote insight and self-awareness within the couple dynamic.
  Arms: Brief Psychoanalytic Couple Therapy (BPCT)
Behavioral: Emotionally Focused Therapy — Emotionally Focused Therapy (EFT) involves 12 weekly online sessions (50 minutes each) focusing on repairing emotional bonds and enhancing attachment security. The intervention targets maladaptive emotional interaction cycles and promotes the expression of primary emotions and attachment needs. Therapists actively guide couples through restructuring emotional responses and rebuilding secure, responsive communication patterns.
  Arms: Emotionally Focused Therapy (EFT)

SUMMARY:
This study compares the effects of two different couple therapy approaches-Brief Psychoanalytic Couple Therapy (BPCT) and Emotionally Focused Therapy (EFT)-on reducing relationship problems and emotional symptoms like depression and anxiety.

Many couples struggle with emotional distance, repeated arguments, and dissatisfaction in their relationships. While EFT is a widely used and research-supported therapy that focuses on rebuilding emotional bonds, BPCT is a less-studied method that aims to help couples understand how early relationship experiences and unconscious patterns affect their current interactions.

The purpose of this study is to find out whether one of these therapies is more effective than the other in improving relationship satisfaction and reducing emotional distress. The study also looks at changes in how people regulate their emotions and how secure they feel in their relationships after therapy.

In this randomized controlled trial, 60 heterosexual couples experiencing relationship distress and symptoms of anxiety or depression will be randomly assigned to one of three groups:

BPCT group - couples receive weekly online therapy focusing on deep emotional and psychological patterns in their relationship.

EFT group - couples receive weekly online therapy focusing on emotional connection and improving communication.

Waitlist control group - couples do not receive therapy during the study but will be offered therapy afterward.

Each therapy lasts 12 weeks, and follow-up assessments will be conducted up to 6 months after therapy ends. Data will be collected before, during, and after treatment using questionnaires that measure relationship satisfaction, depression, anxiety, emotional regulation, and attachment style.

The results of this study will help determine which type of therapy is more beneficial for couples experiencing emotional and relational difficulties and may provide important insights for mental health professionals working with distressed couples.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to compare the clinical efficacy of Brief Psychoanalytic Couple Therapy (BPCT) and Emotionally Focused Therapy (EFT) in reducing relationship distress and associated psychopathological symptoms, including depression, anxiety, and emotional dysregulation. The study also explores secondary outcomes such as changes in adult attachment styles and emotion regulation strategies over time.

While EFT has an established empirical base and is commonly used in clinical practice, BPCT remains underexplored despite its longstanding clinical application. BPCT draws on psychoanalytic principles and focuses on unconscious relational dynamics, early attachment schemas, and defense mechanisms such as projection and transference. EFT, in contrast, is rooted in attachment theory and experiential therapy, emphasizing emotional expression and restructuring maladaptive interaction cycles between partners.

A total of 60 heterosexual couples (n = 120 individuals) experiencing moderate to severe relationship distress-as measured by the Dyadic Adjustment Scale (DAS-32)-and reporting clinically relevant levels of depression and/or anxiety symptoms will be enrolled. Participants will be randomly assigned to one of three arms:

BPCT group (n = 20 couples) - 12 weekly online sessions, each lasting 50 minutes, conducted by trained psychodynamic couple therapists. The focus will be on interpretation of unconscious conflict, symbolic meaning of relational behaviors, and insight into early object relations as they manifest in the couple dynamic.

EFT group (n = 20 couples) - 12 weekly online sessions, also 50 minutes each, delivered by certified EFT therapists. Sessions will center on emotional accessibility, bonding conversations, and reshaping negative emotional cycles.

Waitlist Control group (n = 20 couples) - no therapy during the intervention phase; therapy will be offered following the post-study follow-up assessment.

Assessments will occur at four time points:

Baseline (T0): Full clinical and relational assessments including DAS-32, Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), and the Difficulties in Emotion Regulation Scale (DERS).

Mid-treatment (T1, Week 6): Relationship distress and psychopathology assessments (DAS-32, BDI-II, BAI).

Post-treatment (T2, Week 12): All primary and secondary outcome measures. Follow-up (T3, 6 months after completion): Long-term treatment effects and maintenance of gains.

Statistical analysis will be conducted using repeated measures ANOVA and mixed-effects regression models to account for within-couple dependence and missing data. The Reliable Change Index (RCI) will be used to assess clinically significant change. Between-group effect sizes will also be calculated.

The trial is powered to detect medium effect sizes (Cohen's d = 0.50) with 80% power, accounting for a 20% dropout rate. Therapists will receive supervision to maintain treatment fidelity, and outcome assessors will be blinded to group allocation.

All interventions will be conducted online via secure video conferencing platforms to ensure accessibility and consistency across participants.

This study is expected to contribute significantly to the literature on couple therapy by being the first direct RCT comparison of BPCT and EFT. The findings may inform clinical decision-making regarding the selection of therapeutic models for relational and emotional problems in couples, and potentially promote the integration of psychodynamic and attachment-based frameworks in couple therapy practice.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual couples (both partners must participate)
* Age between 24 and 65 years
* Minimum 2 years of relationship duration
* At least one partner scoring ≤ 30 on the Dyadic Adjustment Scale (DAS-32), indicating clinically significant relationship distress
* At least one partner scoring in the mild, moderate, or severe range on the Beck Depression Inventory-II (BDI-II) or Beck Anxiety Inventory (BAI)

Exclusion Criteria:

* Current participation in individual or couple psychotherapy
* Use of psychiatric medication during the past 3 months
* Presence of severe psychiatric disorders (e.g., psychosis, bipolar disorder)
* History or presence of physical or severe psychological partner violence, assessed via Conflict Tactics Scale (CTS-2)
* Active substance use disorder within the past 6 months

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction (DAS-32) | Baseline, Week 6, Week 12, and 6-month Follow-up
  The Dyadic Adjustment Scale-32 (DAS-32) is a 32-item self-report measure of relationship adjustment. It assesses four subscales: dyadic consensus, satisfaction, cohesion, and affectional expression. Scores range from 0 to 151, with higher scores indicating better relationship quality. A score below 100 indicates relationship distress. Changes will be assessed across the four time points to evaluate therapeutic impact.
Change in Depressive Symptoms (BDI-II) | Baseline, Week 6, Week 12, and 6-month Follow-up
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report questionnaire measuring the severity of depressive symptoms. Scores range from 0 to 63. Scores between 14-19 reflect mild depression, 20-28 moderate, and 29-63 severe. Higher scores indicate greater severity. The change in BDI-II scores will be used to assess symptom improvement.
Change in Anxiety Symptoms (BAI) | Baseline, Week 6, Week 12, and 6-month Follow-up
  The Beck Anxiety Inventory (BAI) is a 21-item self-report inventory that measures the severity of anxiety symptoms. Scores range from 0 to 63, with scores above 16 indicating clinically significant anxiety. Higher scores indicate more severe anxiety. Changes in BAI scores will track anxiety symptom reduction.
Change in Emotion Dysregulation (DERS) | Baseline, Week 12, and 6-month Follow-up
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item measure assessing six dimensions of emotion regulation: nonacceptance, goals, impulse, awareness, strategies, and clarity. Total scores range from 36 to 180, with higher scores indicating more difficulties in emotion regulation. Changes in total scores across time points will be evaluated.

SECONDARY OUTCOMES:
Change in Adult Attachment Style (AAS) | Baseline, Week 12, and 6-month Follow-up
  The Couples Satisfaction Index-4 (CSI-4) is a brief, 4-item scale designed to assess global relationship satisfaction. Responses are based on Likert-type items. Scores range from 0 to 21, with higher scores reflecting greater satisfaction. The CSI-4 has demonstrated strong internal consistency and criterion validity. Changes in CSI-4 scores will be used as a secondary index of intervention effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Gökben Hızlı Sayar, Professor, Study Chair — Üsküdar University; Metin Çınaroğlu, Phd, Study Director — İstanbul Nişantaşı University
Locations (1):
- Beykoz University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures-including DAS-32, BDI-II, BAI, DERS, CSI-4, and AAS scores-will be made available for secondary analysis upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD and supporting documentation will be available beginning 6 months after the publication of primary results and for up to 5 years upon reasonable request.
Access Criteria: Qualified researchers affiliated with academic or nonprofit institutions may request access to de-identified data for ethically approved studies. Requests will be reviewed by the principal investigator. Data will be shared via secure email or institutional repository upon approval and signed data use agreement.